CLINICAL TRIAL: NCT01400841
Title: A Prospective, Non-randomized, Multi-center Trial to Evaluate the Safety and Effectiveness of the HAART Model 300 Annuloplasty Ring When Used to Surgically Repair a Leaking Aortic Valve Using a 3-D Intra-annular Mounting Frame
Brief Title: HAART Model 300 Annuloplasty Ring
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biostable Science & Engineering (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BSE 300; TP-01-013 (Other: Biostable Science & Engineering, Inc); TP-01-023 (Other: Biostable Science & Engineering, Inc)
Record Dates: First submitted 2011-07-21; First posted 2011-07-22 (Estimated); Results first posted 2016-11-22 (Estimated); Last update posted 2017-01-13 (Estimated); Status verified 2016-11

CONDITIONS: Aortic Regurgitation
Keywords: Aortic Insufficiency, Aortic Regurgitation, Aortic Valve Repair
MeSH Terms: conditions — Aortic Valve Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- HAART 300 Annuloplasty Device (Experimental): Implantation of HAART 300 Annuloplasty Device for aortic valve repair
  Interventions: Device: HAART 300 Annuloplasty Device

INTERVENTIONS:
Device: HAART 300 Annuloplasty Device — Implantation of device for aortic valve repair

SUMMARY:
This investigation is a prospective, non-randomized, multi-center trial to evaluate the safety and effectiveness of the HAART model 300 annuloplasty ring when used to surgically repair a leaking aortic valve using a 3-D intra-annular mounting frame

DETAILED DESCRIPTION:
Aortic Regurgitation, (also known as Aortic Insufficiency; AI), is the failure of the aortic valve to close completely during diastole which causes blood to flow from the aorta back into the left ventricle. Aortic Regurgitation (AR) is a frequent cause of both disability and death due to congestive heart failure, primarily in individuals forty or older, but can also occur in younger populations.

Traditionally management of aortic regurgitation has been by aortic valve replacement, however, as has been observed in patients who have had mitral valve repair, the option of maintaining ones native aortic valve versus a replacement, either bioprosthetic or mechanical, can have added multiple benefits. The advantage of repair is the avoidance of prosthetic valve-related complications with bioprosthetic valves over 10-15 years or the need for anticoagulation with mechanical valves and the related problems of this therapy. Therefore, potentially aortic valve repair is a good option for patients with AR or AI.

ELIGIBILITY:
Inclusion Criteria:

* The subject is 50 years old or older
* The subject has a tricuspid aortic valve morphology
* Patients with documented severe aortic insufficiency with aortic annular dilation without severe concomitant aortic stenosis
* Patients referred to center for documented moderate to severe Chronic aortic regurgitation (AR) associated with annular dilatation with or without cusp prolapse of one, two, or all three leaflets
* Patients with or without Sinotubular Junction (STJ) dilatation or aortic root aneurysms
* Patients who are free of coronary disease or those with evidence of minor stable (1-2 vessel) coronary disease
* Subject is willing to comply with specified follow-up evaluations, including transesophageal echocardiography if there are inadequate images by transthoracic echocardiography (TTE) to assess the aortic valve
* The subject has signed the written informed consent
* The subject agrees to return for all follow-up evaluations for the duration of the study (i.e. geographically stable
* The subject is New York Hospital Association (NYHA) class II or III

Exclusion Criteria:

* The subject has preexisting valve prosthesis in the atrial, the mitral, pulmonary, and/or tricuspid position
* The subject requires an additional valve replacement
* The subject's aortic valve morphology is not tricuspid
* The subject has active endocarditis
* Heavily calcified valves
* Valvular retraction with severely reduced mobility
* The subject has mixed stenosis and regurgitation of the aortic valve with predominant stenosis
* The subject requires a repair of the mitral or tricuspid valve with the use of an annuloplasty device
* Leukopenia
* Acute anemia (Hb < 9mg%)
* Platelet count <100,000 cell/mm3
* Need for emergency surgery for any reason
* History of bleeding diathesis or coagulopathy or the subject refuses blood transfusions
* Active infection requiring antibiotic therapy (if temporary illness, subjects may enroll 4 weeks after discontinuation of antibiotics)
* Subjects in whom transesophageal echocardiography (TEE) is contraindicated
* Non elective presentation
* Low Ejection Fraction (EF) EF < 40%
* Life expectancy < 1 year
* Rheumatic disease
* The subject has severe leaflet fenestration or leaflets damaged by endocarditis
* The subject is or will be participating in a concomitant research study of an investigational product or has participated in such a study within the 30 days prior to screening
* The subject is a minor, an illicit drug user, alcohol abuser, prisoner, institutionalized, or is unable to give informed consent
* The subject is pregnant or lactating
* This patient will not agree to return to the implant center for the required number of follow-up visits or is geographically unavailable for follow-up
* The subject has not signed and dated the study informed consent
* Recent (within 6 months) cerebrovascular accident (CVA) or transient ischemic attack (TIA)
* Myocardial infarction (MI) within one month of trial inclusion
* Have a known intolerance to titanium or polyester
* Sole therapy for correction for patients with aortic root aneurysm
* Subjects requiring simultaneous cardiac procedures
* The subject has asymptomatic AR and a left ventricular ejection fraction (LVEF) > 50%

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2012-01; Primary Completion 2013-04 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christof Stamm, M.D., Principal Investigator — German Heart Institute
Locations (4):
- University Hospital Gasthuisberg, Leuven, Belgium
- Institut klinicke a experimantalni mediciny, Prague, Czechia
- Germany (2):
  - German Heart Institute, Berlin
  - German Heart Center Munich, Munich

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Mazzitelli D, Fischlein T, Rankin JS, Choi YH, Stamm C, Pfeiffer S, Pirk J, Detter C, Kroll J, Beyersdorf F, Griffin CD, Shrestha M, Nobauer C, Crooke PS, Schreiber C, Lange R. Geometric ring annuloplasty as an adjunct to aortic valve repair: clinical investigation of the HAART 300 device. Eur J Cardiothorac Surg. 2016 Mar;49(3):987-93. doi: 10.1093/ejcts/ezv234. Epub 2015 Jul 8. PMID 26156945
- [Derived] Mazzitelli D, Stamm C, Rankin JS, Pfeiffer S, Fischlein T, Pirk J, Choi YH, Detter C, Kroll J, Beyersdorf F, Shrestha M, Schreiber C, Lange R. Leaflet reconstructive techniques for aortic valve repair. Ann Thorac Surg. 2014 Dec;98(6):2053-60. doi: 10.1016/j.athoracsur.2014.06.052. Epub 2014 Dec 1. PMID 25468084
- [Derived] Mazzitelli D, Stamm C, Rankin JS, Nobauer C, Pirk J, Meuris B, Crooke PS, Wagner A, Beavan LA, Griffin CD, Powers D, Nasseri B, Schreiber C, Hetzer R, Lange R. Hemodynamic outcomes of geometric ring annuloplasty for aortic valve repair: a 4-center pilot trial. J Thorac Cardiovasc Surg. 2014 Jul;148(1):168-75. doi: 10.1016/j.jtcvs.2013.08.031. Epub 2013 Oct 8. PMID 24113022
- [Derived] Mazzitelli D, Nobauer C, Rankin JS, Badiu CC, Dorfmeister M, Crooke PS, Wagner A, Schreiber C, Lange R. Early results of a novel technique for ring-reinforced aortic valve and root restoration. Eur J Cardiothorac Surg. 2014 Mar;45(3):426-30. doi: 10.1093/ejcts/ezt407. Epub 2013 Aug 19. PMID 23959743

RESULTS

PARTICIPANT FLOW:
Period: Initial Study Phase (6 Months)
Arm/Group | HAART 300 Annuloplasty Device
Started | 16 (2 of the 18 consented subjects did not receive the device)
Completed | 15
Not Completed | 1
Not completed — Death | 1
Period: Extended Study Phase (2 Years)
Arm/Group | HAART 300 Annuloplasty Device
Started | 13 (1 subject refused further participation 1 subject death prior to agreeing to extended follow-up)
Completed | 11
Not Completed | 2
Not completed — Adverse Event | 2

BASELINE CHARACTERISTICS:
Arm/Group | HAART 300 Annuloplasty Device
Number analyzed (Participants) | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.1 (9.3)
Gender [Count of Participants; unit: Participants]
  Female | 3
  Male | 13
Region of Enrollment [Number; unit: participants]
  Czech Republic | 2
  Belgium | 1
  Germany | 13
Aortic Valvular Regurgitation [Number; unit: participants] — Grade assigned to degree of aortic regurgitation determined by core laboratory analysis of echocardiogram: 0=None/trace, 1+=Mild, 2+=Moderate, 3+=Moderate-to-Severe, 4+=Severe
  participants
    0 | 0
    1+ | 0
    2+ | 6
    3+ | 7
    4+ | 3
NYHA Classification [Number; unit: participants] — New York Heart Association Functional Capacity
  Class I: no limitation of activity. Ordinary activity - no undue fatigue, palpitation, dyspnea, or anginal pain.
  Class II: slight limitation of activity. Comfortable at rest. Ordinary activity - fatigue, palpitation, dyspnea, or anginal pain.
  Class III: marked limitation of activity. Comfortable at rest. Less than ordinary activity - fatigue, palpitation, dyspnea, or anginal pain.
  Class IV: no activity without discomfort. Symptoms of heart failure or the anginal syndrome may be present even at rest. Increased discomfort upon activity.
  participants
    I | 0
    II | 10
    III | 6
    IV | 0
Peak gradient [Mean (Standard Deviation); unit: mm Hg] — Echocardiographic parameter determined by core laboratory. n=14 (2 unavailable or not evaluable)
  mm Hg | 13.3 (6.2)
Mean gradient [Mean (Standard Deviation); unit: mm Hg] — Echocardiographic parameter determined by core laboratory. n=14 (2 unavailable or not evaluable)
  mm Hg | 6.8 (3.0)
Left ventricular (LV) mass [Mean (Standard Deviation); unit: g] — Left ventricular mass. Echocardiographic parameter determined by core laboratory. n=11 (5 unavailable or not evaluable)
  g | 260.0 (57.1)
Left ventricular internal dimension (LVID) diastole [Mean (Standard Deviation); unit: cm] — Left ventricular internal dimension. Echocardiographic parameter determined by core laboratory. n=11 (5 unavailable or not evaluable)
  cm | 5.44 (0.60)
LVID systole [Mean (Standard Deviation); unit: cm] — Left ventricular internal dimension. Echocardiographic parameter determined by core laboratory. n=7 (9 unavailable or not evaluable)
  cm | 4.09 (0.76)
LV diastolic volume [Mean (Standard Deviation); unit: ml] — Left ventricular diastolic volume. Echocardiographic parameter determined by core laboratory. n=10 (6 unavailable or not evaluable)
  ml | 180.7 (50.2)
LV systolic volume [Mean (Standard Deviation); unit: ml] — Left ventricular systolic volume. Echocardiographic parameter determined by core laboratory. n=10 (6 unavailable or not evaluable)
  ml | 84.7 (25.4)
Left ventricular ejection fraction (LVEF) [Mean (Standard Deviation); unit: %] — Left ventricular ejection fraction. Echocardiographic parameter determined by core laboratory. n=10 (6 unavailable or not evaluable)
  % | 53.2 (6.7)
Cardiac output [Mean (Standard Deviation); unit: l/min] — Echocardiographic parameter determined by core laboratory. n=9 (7 unavailable or not evaluable)
  l/min | 6.77 (1.60)
Cardiac index [Mean (Standard Deviation); unit: l/min/m^2] — Cardiac index is the cardiac output divided by body surface area. n=9 (7 unavailable or not evaluable)
  l/min/m^2 | 3.41 (0.90)

OUTCOME MEASURES:

1. Primary Outcome: Primary Safety Outcome Measure: Event-free Survival
Description: Event-free survival is defined as survival free from device-related death
Time Frame: 1 month postprocedure
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | HAART 300 Annuloplasty Device
Number analyzed (Participants) | 16
percentage of participants | 100 [79.4 to 100]

2. Primary Outcome: Primary Safety Outcome Measure: Event-free Survival
Description: Event-free survival is defined as survival free from device-related death
Time Frame: 2 years postprocedure (extended follow-up)
Population: Extended follow-up participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | HAART 300 Annuloplasty Device
Number analyzed (Participants) | 13
percentage of participants | 100 [75.3 to 100]

3. Primary Outcome: Primary Efficacy Outcome Measure: Aortic Valvular Regurgitation at 6 Months Postprocedure
Description: Aortic valvular regurgitation assessed by transthoracic echocardiography and graded as None/Trace (0), Mild (1+), Moderate (2+), Moderate-to-Severe (3+), or Severe (4+)
Time Frame: 6 months postprocedure
Measure: Number; unit: participants
Arm/Group | HAART 300 Annuloplasty Device
Number analyzed (Participants) | 15
participants
  0 | 2
  1+ | 9
  2+ | 3
  3+ | 1
  4+ | 0

4. Primary Outcome: Primary Efficacy Outcome Measure: Aortic Valvular Regurgitation at 2 Years Postprocedure
Description: as for outcome 3
Time Frame: 2 years postprocedure (extended follow-up)
Measure: Number; unit: participants
Arm/Group | HAART 300 Annuloplasty Device
Number analyzed (Participants) | 11
participants
  0 | 2
  1+ | 7
  2+ | 2
  3+ | 0
  4+ | 0

5. Secondary Outcome: Implant Procedure Success
Description: Success is defined as the absence of specified adverse events evaluated through discharge or 14 days after the procedure:
  * Aortic annular dissection, rupture, or leaflet damage
  * Paravalvular leak > +2 or requiring intervention
  * Mitral valve impingement due to implant
  * implant dehiscence/migration into aorta
  * implant dehiscence/migration into left ventricle
  * Hemodynamics requiring intervention
  * Other adverse event resulting in reoperation, explantation, or permanent disability.
Time Frame: discharge or 14 days postprocedure, whichever comes first
Measure: Number (95% Confidence Interval); unit: percentage of implant procedures
Arm/Group | HAART 300 Annuloplasty Device
Number analyzed (Participants) | 16
percentage of implant procedures | 100 [79.4 to 100]

6. Secondary Outcome: Implant Procedure Success
Description: as for outcome 5
Time Frame: 2 years postprocedure (extended follow-up)
Measure: Number (95% Confidence Interval); unit: percentage of implant procedures
Arm/Group | HAART 300 Annuloplasty Device
Number analyzed (Participants) | 16
percentage of implant procedures | 87.5 [61.6 to 98.4]

7. Secondary Outcome: Actuarial Freedom From Clinical Cardiovascular Events
Description: Freedom from specified clinical cardiovascular events 1 month postprocedure:
  * Device-related mortality
  * Complete heart block
  * Structural device failure
  * Endocarditis
  * Periprosthetic leak or dehiscence
  * Thromboembolism
  * Bleeding Event
  * Native Valve Deterioration
  * Valve Thrombosis
  * Hemolysis
  * Reoperation and explant at 1 month
Time Frame: 1 month postprocedure
Measure: Number (95% Confidence Interval); unit: percentage of implant procedures
Arm/Group | HAART 300 Annuloplasty Device
Number analyzed (Participants) | 16
percentage of implant procedures | 100 [79.4 to 100]

8. Secondary Outcome: Actuarial Freedom From Clinical Cardiovascular Events
Description: Freedom from specified clinical cardiovascular events 2 years postprocedure:
  * Device-related mortality
  * Complete heart block
  * Structural device failure
  * Endocarditis
  * Periprosthetic leak or dehiscence
  * Thromboembolism
  * Bleeding Event
  * Native Valve Deterioration
  * Valve Thrombosis
  * Hemolysis
  * Reoperation and explant at 2 years
Time Frame: 2 years postprocedure
Measure: Number (95% Confidence Interval); unit: percentage of implant procedures
Arm/Group | HAART 300 Annuloplasty Device
Number analyzed (Participants) | 16
percentage of implant procedures | 81.5 [53.4 to 100]

9. Secondary Outcome: Event-free Survival
Description: Event-free survival is defined as survival free from device-related death
Time Frame: 6 months postprocedure
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | HAART 300 Annuloplasty Device
Number analyzed (Participants) | 16
percentage of participants | 100 [79.4 to 100]

10. Secondary Outcome: New York Heart Association (NYHA) Functional Capacity Classification
Description: Four classes describing the effect of cardiac disease on physical activity: Class I - disease does not limit activity; Class II - slight limitation; Class III - marked limitation; Class IV - inability to carry out any physical activity without discomfort
Time Frame: 6 months postprocedure
Population: NYHA evaluation not done on 1 of 15 participants
Measure: Number; unit: participants
Arm/Group | HAART 300 Annuloplasty Device
Number analyzed (Participants) | 14
participants
  I | 11
  II | 3
  III | 0
  IV | 0

11. Secondary Outcome: New York Heart Association (NYHA) Functional Capacity Classification
Description: as for outcome 10
Time Frame: 2 years postprocedure (extended follow-up)
Measure: Number; unit: participants
Arm/Group | HAART 300 Annuloplasty Device
Number analyzed (Participants) | 11
participants
  I | 8
  II | 3
  III | 0
  IV | 0

12. Secondary Outcome: Peak Gradient - Change From Baseline
Description: Transthoracic echocardiography parameter
Time Frame: Baseline, 6 months postprocedure
Population: Baseline measure not available for 1 of 15 participants.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | HAART 300 Annuloplasty Device
Number analyzed (Participants) | 14
mm Hg | 4.9 (5.6)

13. Secondary Outcome: Peak Gradient - Change From Baseline
Description: Transthoracic echocardiography parameter
Time Frame: Baseline, 2 years postprocedure (extended follow-up)
Population: Baseline measure not available for 1 of 11 participants.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | HAART 300 Annuloplasty Device
Number analyzed (Participants) | 10
mm Hg | 10.1 (9.4)

14. Secondary Outcome: Mean Gradient - Change From Baseline
Description: Transthoracic echocardiography parameter
Time Frame: Baseline, 6 months postprocedure
Population: Baseline measure not available for 1 of 15 participants.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | HAART 300 Annuloplasty Device
Number analyzed (Participants) | 14
mm Hg | 2.6 (2.7)

15. Secondary Outcome: Mean Gradient - Change From Baseline
Description: Transthoracic echocardiography parameter
Time Frame: Baseline, 2 years postprocedure (extended follow-up)
Population: Baseline measure not available for 1 of 11 participants.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | HAART 300 Annuloplasty Device
Number analyzed (Participants) | 10
mm Hg | 4.8 (4.8)

16. Secondary Outcome: LV Mass - Change From Baseline
Description: Left ventricular mass. Transthoracic echocardiography parameter.
Time Frame: Baseline, 6 months postprocedure
Population: Both baseline and 6-month measure available for 8 of 15 participants
Measure: Mean (Standard Deviation); unit: g
Arm/Group | HAART 300 Annuloplasty Device
Number analyzed (Participants) | 8
g | -53.4 (57.1)

17. Secondary Outcome: LV Mass - Change From Baseline
Description: Left ventricular mass. Transthoracic echocardiography parameter.
Time Frame: Baseline, 2 years postprocedure (extended follow-up)
Population: Both baseline and 2-year measure available for 6 of 11 participants.
Measure: Mean (Standard Deviation); unit: g
Arm/Group | HAART 300 Annuloplasty Device
Number analyzed (Participants) | 6
g | -23.3 (72.0)

18. Secondary Outcome: LVID Diastole - Change From Baseline
Description: Left ventricular internal dimension. Transthoracic echocardiography parameter.
Time Frame: Baseline, 6 months postprocedure
Population: Both baseline and 6-month measure available for 8 of 15 participants.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | HAART 300 Annuloplasty Device
Number analyzed (Participants) | 8
cm | -0.52 (0.61)

19. Secondary Outcome: LVID Diastole - Change From Baseline
Description: Left ventricular internal dimension. Transthoracic echocardiography parameter.
Time Frame: Baseline, 2 years postprocedure (extended follow-up)
Population: Both baseline and 2-year measure available for 7 of 11 participants.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | HAART 300 Annuloplasty Device
Number analyzed (Participants) | 7
cm | -0.33 (0.82)

20. Secondary Outcome: LVID Systole - Change From Baseline
Description: Left ventricular internal dimension. Transthoracic echocardiography parameter.
Time Frame: Baseline, 6 months postprocedure
Population: Both baseline and 6-month measure available for 5 of 15 participants.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | HAART 300 Annuloplasty Device
Number analyzed (Participants) | 5
cm | -0.75 (0.68)

21. Secondary Outcome: LVID Systole - Change From Baseline
Description: Left ventricular internal dimension. Transthoracic echocardiography parameter.
Time Frame: Baseline, 2 years postprocedure (extended follow-up)
Population: Both baseline and 2-year measure available for 3 of 11 participants.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | HAART 300 Annuloplasty Device
Number analyzed (Participants) | 3
cm | 0.03 (1.09)

22. Secondary Outcome: LV Diastolic Volume - Change From Baseline
Description: Left ventricular diastolic volume. Transthoracic echocardiography parameter.
Time Frame: Baseline, 6 months postprocedure
Population: Both baseline and 6-month measure available for 7 of 15 participants.
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | HAART 300 Annuloplasty Device
Number analyzed (Participants) | 7
ml | -49.9 (64.2)

23. Secondary Outcome: LV Diastolic Volume - Change From Baseline
Description: Left ventricular diastolic volume. Transthoracic echocardiography parameter.
Time Frame: Baseline, 2 years postprocedure (extended follow-up)
Population: Both baseline and 2-year measure available for 5 of 11 participants.
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | HAART 300 Annuloplasty Device
Number analyzed (Participants) | 5
ml | -75.4 (74.3)

24. Secondary Outcome: LV Systolic Volume - Change From Baseline
Description: Left ventricular systolic volume. Transthoracic echocardiography parameter.
Time Frame: Baseline, 6 months postprocedure
Population: Both baseline and 6-month measure available for 7 of 15 participants.
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | HAART 300 Annuloplasty Device
Number analyzed (Participants) | 7
ml | -30.6 (30.2)

25. Secondary Outcome: LV Systolic Volume - Change From Baseline
Description: Left ventricular systolic volume. Transthoracic echocardiography parameter.
Time Frame: Baseline, 2 years postprocedure (extended follow-up)
Population: Both baseline and 2-year measure available for 5 of 11 participants.
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | HAART 300 Annuloplasty Device
Number analyzed (Participants) | 5
ml | -48.4 (38.2)

26. Secondary Outcome: LVEF - Change From Baseline
Description: Left ventricular ejection fraction. Transthoracic echocardiography parameter.
Time Frame: Baseline, 6 months postprocedure
Population: Both baseline and 6-month measure available for 7 of 15 participants.
Measure: Mean (Standard Deviation); unit: percentage of blood volume
Arm/Group | HAART 300 Annuloplasty Device
Number analyzed (Participants) | 7
percentage of blood volume | 5.13 (6.53)

27. Secondary Outcome: LVEF - Change From Baseline
Description: Left ventricular ejection fraction. Transthoracic echocardiography parameter.
Time Frame: Baseline, 2 years postprocedure (extended follow-up)
Population: Both baseline and 2-year measure available for 5 of 11 participants.
Measure: Mean (Standard Deviation); unit: percentage of blood volume
Arm/Group | HAART 300 Annuloplasty Device
Number analyzed (Participants) | 5
percentage of blood volume | 12.20 (9.57)

28. Secondary Outcome: Cardiac Output - Change From Baseline
Description: Stroke volume x heart rate. Transthoracic echocardiography parameter.
Time Frame: Baseline, 6 months postprocedure
Population: Both baseline and 6-month measure available for 7 of 15 participants.
Measure: Mean (Standard Deviation); unit: l/min
Arm/Group | HAART 300 Annuloplasty Device
Number analyzed (Participants) | 7
l/min | -0.73 (1.55)

29. Secondary Outcome: Cardiac Output - Change From Baseline
Description: Stroke volume x heart rate. Transthoracic echocardiography parameter.
Time Frame: Baseline, 2 years postprocedure (extended follow-up)
Population: Both baseline and 2-year measure available for 5 of 11 participants.
Measure: Mean (Standard Deviation); unit: l/min
Arm/Group | HAART 300 Annuloplasty Device
Number analyzed (Participants) | 5
l/min | -0.36 (0.34)

30. Secondary Outcome: Cardiac Index - Change From Baseline
Description: Hemodynamic parameter computed as cardiac output divided by body surface area
Time Frame: Baseline, 6 months postprocedure
Population: Both baseline and 6-month measure available for 7 of 15 participants.
Measure: Mean (Standard Deviation); unit: l/min/m^2
Arm/Group | HAART 300 Annuloplasty Device
Number analyzed (Participants) | 7
l/min/m^2 | -0.40 (0.80)

31. Secondary Outcome: Cardiac Index - Change From Baseline
Description: Hemodynamic parameter computed as cardiac output divided by body surface area
Time Frame: Baseline, 2 years postprocedure (extended follow-up)
Population: Both baseline and 2-year measure available for 5 of 11 participants.
Measure: Mean (Standard Deviation); unit: l/min/m^2
Arm/Group | HAART 300 Annuloplasty Device
Number analyzed (Participants) | 5
l/min/m^2 | -0.22 (0.18)

ADVERSE EVENTS:
Time Frame: Through 6 months for 16 participant receiving the implant and through 2 years for 13 of the 16 participants in extended follow-up
Arm/Group | HAART 300 Annuloplasty Device
Serious Adverse Events (participants affected / at risk) | 8/16
Other Adverse Events (participants affected / at risk) | 15/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HAART 300 Annuloplasty Device (N=16)
aortic insufficiency (Cardiac disorders) | 2 (2)
arrhythmia (Cardiac disorders) | 1 (1)
syncope (Cardiac disorders) | 2 (2)
GI bleeding (Gastrointestinal disorders) | 1 (1)
central venous catheter infection (Infections and infestations) | 1 (1)
primary coxarthrosis left (Musculoskeletal and connective tissue disorders) | 1 (1)
radial fracture (Musculoskeletal and connective tissue disorders) | 1 (1)
choreiform movement disorder (Nervous system disorders) | 1 (1)
postop delirium (Nervous system disorders) | 1 (1)
urinary tract infection (Renal and urinary disorders) | 1 (1)
subcutaneous emphysema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HAART 300 Annuloplasty Device (N=16)
anemia (Blood and lymphatic system disorders) | 1 (1)
enhanced plasma free hemoglobin value (Blood and lymphatic system disorders) | 3 (3)
arrhythmia (Cardiac disorders) | 9 (9)
conduction defects (Cardiac disorders) | 1 (1)
intramural aortic hematoma (Cardiac disorders) | 1 (1)
pericardial effusion (Cardiac disorders) | 6 (6)
chest pain (Injury, poisoning and procedural complications) | 1 (1)
cicatrical hernia (Injury, poisoning and procedural complications) | 1 (1)
reddening of wound (Injury, poisoning and procedural complications) | 1 (1)
arthrosis left knee (Musculoskeletal and connective tissue disorders) | 1 (1)
back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
hip pain (Musculoskeletal and connective tissue disorders) | 1 (1)
leg pain (Musculoskeletal and connective tissue disorders) | 1 (1)
thoracal pain (Musculoskeletal and connective tissue disorders) | 1 (1)
pulmonary mass (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
flickering in the eyes (Nervous system disorders) | 1 (1)
numbness of left little finger (Nervous system disorders) | 1 (1)
postoperative delirium (Nervous system disorders) | 1 (1)
symptomatic transitory psychotic syndrome (Nervous system disorders) | 1 (1)
cystitis (Renal and urinary disorders) | 2 (2)
hematuria (Renal and urinary disorders) | 1 (1)
atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
flu with fever (Respiratory, thoracic and mediastinal disorders) | 1 (1)
mild cold (Respiratory, thoracic and mediastinal disorders) | 1 (1)
pleural effusion (Respiratory, thoracic and mediastinal disorders) | 7 (7)
pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
clavus (Skin and subcutaneous tissue disorders) | 1 (1)
thrombophlebitis (Vascular disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publication by the investigator was not allowed until completion of the trial. All proposed publications must be cleared by unanimous vote of a publication committee consisting of the sponsor and representatives of the study investigators. Publication materials must be submitted for review at least 60 day in advance of publication. The Sponsor may embargo publication for 60 additional days to allow for patent filing or may prevent publication if filling of such application would be premature.